CLINICAL TRIAL: NCT03769935
Title: Preliminary Study of Maintenance Therapy for Patients With Extensive Stage of Small-cell Lung Cancer
Brief Title: Maintenance Therapy for Small-cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QingdaoCH2018-12-02
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Progression Free Survival
MeSH Terms: interventions — Cisplatin; Etoposide; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental arm (Experimental): cisplatin 75 mg/m2, iv day1, Etoposide: 60 mg/m2 IV day 1-5, every 21 days for up to 4-6 cycles.
  S1 25 mg/m2 oral, everyday until progression disease
  Interventions: Drug: cis Platinum, etoposide, S1
- active comparator (Active Comparator): cisplatin 75 mg/m2, iv day1, Etoposide: 60 mg/m2 IV day 1-5, every 21 days for up to 4-6 cycles.
  Interventions: Drug: cis Platinum, etoposide, S1

INTERVENTIONS:
Drug: cis Platinum, etoposide, S1 — cisplatin 75 mg/m2, iv day1, Etoposide: 60 mg/m2 IV day 1-5, every 21 days for up to 4-6 cycles.
  S1 25 mg/m2 oral, everyday until progression disease

SUMMARY:
This study involves patients treated with cisplatin and etoposide (induction therapy), followed by treatment with a drug called S1 (maintenance therapy). The main purpose of this study is to determine if this type of treatment will delay the growth of the tumor and if so, for how long. The primary endpoint is progression free survival and second endpoints are toxicities, overall survival.

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) accounts for about 20% of lung cancer, has a high degree of malignancy, short doubling time, early and widespread metastasis, is sensitive to chemotherapy and radiotherapy, and has a high initial response rate, but is prone to secondary drug resistance and relapse. The treatment is mainly based on systemic chemotherapy, and if maintenance therapy with S1 after standard EP regimen induction therapy could prolong progression free survival.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histopathologically confirmed patients with extensive small cell lung cancer; 2. Karnofsky performance status ≥60; 3. At least one lesion that can measured by CT; 4. Expected to survive for at least 3 months; 5. Peripheral blood and liver and kidney function within the following allowable range (tested within 7 days before treatment); 6. White blood cell (WBC) ≥3.0×109/L or Neutrophils (ANC) ≥1.5×109/L; Hemoglobin (HGB) ≥80 g/L；Platelet (PLT) ≥100×109/L; 7. Liver transaminases（AST/ALT）<3.0 times the normal range limit; Total bilirubin（TBIL）<1.5 times the normal range limit; Creatinine（CREAT）<1.5 times the normal range limit; 8. Patients of childbearing age (including female and male patients' partner) must take effective contraception methods; Signed informed consent 9. Must be able to swallow tablets

Exclusion Criteria:

* 1. Limited stage disease 2. Metastastic meningitis, spinal compression, Tumor to main vesicular less than 5mm 3. Other pathological types of tumor except for small cell lung cancer; 4. Patients with a history of severe allergies or allergies; 5. Pregnancy or breastfeeding women; 6. Patients who have previously participated in other clinical trials and have not yet terminated the trial; 7. Patients who have acute infection that difficult to control; 8. Subjects with difficulties in swallowing or known drug malabsorption.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
The progression-free survival in this population of patients | 2.5 years
  The progression-free survival of the enrolled patients from start the combination treatment with cisplatin, etoposide and S1

SECONDARY OUTCOMES:
Percentage of Participants Experiencing an Adverse Event (AE) | 2.5 years
  Adverse events were recorded and classified from start the treatment by grade according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0
The overall survival in this population of patients. | 2.5 years
  The overall survival of the enrolled patients from start the combination from start the combination treatment with cisplatin, etoposide and S1

CONTACTS AND LOCATIONS:
Locations (1):
- Qingdao Central Hospital, Qingdao Cancer Hospital, Qingdao, Shandong, China